CLINICAL TRIAL: NCT00828126
Title: PET-CT in the Management of Patients With Stage III Or IV Metastatic Melanoma Considered Candidates for Surgery: Evaluation of Additive Value Following Conventional Imaging
Brief Title: PET-CT in the Management of Patients With Stage III or IV Metastatic Melanoma
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0478
Record Dates: First submitted 2009-01-13; First posted 2009-01-23 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Melanoma
Keywords: Metastatic Melanoma; AJCC Stage III Melanoma; AJCC stage IV Melanoma; PET-CT; Positron Emission Tomography-Computed Tomography; Contrast-enhanced Computed Tomography Scan; CT; Conventional Imaging; False Positive Rate; Fluorodeoxyglucose; FDG; Surgery
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET-CT Scan
  Interventions: Procedure: PET-CT Scan

INTERVENTIONS:
Procedure: PET-CT Scan — Positron emission tomography-computed tomography (PET-CT) scan performed within 30 days of contrast-enhanced CT.
  Other Names: PET-CT

SUMMARY:
The goal of this clinical research study is to learn how often using a positron emission tomography-computed tomography (PET-CT) scan in addition to a standard computed tomography (CT) scan will change the surgical plan in patients with metastatic melanoma.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will have a PET-CT scan performed. The picture produced by this scan will be compared to a standard CT scan to see if any additional tumors can be located. If the study doctor thinks that additional tumors are present, a biopsy may need to be performed to check the status of the tumors. The type of biopsy will depend on where the tumor(s) are located on the body. If a biopsy is performed, you will sign a separate consent.

Screening Tests:

Women who decide to take part in this study will be asked if they think they might be pregnant at the start of the study. Women who are unsure if they may be pregnant or think that they may be pregnant must have a negative blood (about 1 teaspoon) pregnancy test.

PET-CT Scan Procedure:

Before the PET-CT scan is performed, you will be asked to avoid stressful exercise for 24 hours. Starting about 12 hours before the scan, you should eat a high protein diet and limit the amount of carbohydrates you eat. Starting about 6 hours before the scan, you should not eat or drink anything other than water (fast) until after the scan is done. You may continue to take prescribed drugs with water during the fasting period.

On the day of the PET-CT scan, you should wear comfortable clothing, preferably without metal buttons and/or zippers. You will be asked to remove any metallic objects you have when you arrive at the PET-CT Center.

* Blood (a few drops from the fingertip) will be collected to check your blood sugar levels.
* A radioactive sugar solution, called fluorodeoxyglucose (FDG), will be given through a needle in a vein of your arm. The injection will last about 5 minutes. Following the FDG injection, you will rest for about 1 hour to allow the FDG to move throughout the body. You will then be asked to urinate before the scan is performed.

You will lie flat on your back on the scanner table. The table will move slowly in and out of a donut-shaped machine called the PET-CT scanner. This scanner creates a picture that shows the FDG in the tumor(s) and organs. The scan takes about 45-60 minutes. You will need to lie as still as possible while the scan is being performed.

Length of Study:

Your participation on this study will be over after PET-CT scan has been completed.

Follow-Up Visits:

As a part of your standard of care, your primary care physician may order additional imaging after your completion of this study for follow-up purposes. The study doctor will review these images to compare them with the PET-CT images. The study doctors will also review the results of any biopsies you may have had as a result of PET-CT findings.

This is an investigational study. PET-CT and CT scans are FDA approved and commercially available. The PET-CT component of this study is investigational because it is being done within a certain timeframe (within 30 days after your CT scan) instead of at the timeframe your doctor would normally decide.

Up to 150 patients will take part in this study. All will be enrolled at M. D. Anderson Cancer Center (MDACC).

ELIGIBILITY:
Inclusion Criteria:

1. AJCC Stage III melanoma with clinically evident (macroscopic) disease, either by physical examination or on conventional imaging, or AJCC stage IV melanoma with metastatic site(s) considered surgically resectable. The initial decision regarding surgical candidacy should be made by surgical oncologist. Patients with indeterminate CT findings that are larger than 1 cm outside of the field of the potential surgery will be also included.
2. Contrast- enhanced CT of chest, abdomen and pelvis performed either at MDACC or outside of the institution should indicate surgical candidacy. Outside CT imaging studies should be of acceptable quality, as determined by the evaluating radiologist. PET-CT per protocol must be performed within 30 days from the contrast-enhanced CT.
3. 3. Age >/= 18. All minor patients will be excluded to avoid excessive radiation dose. There is data suggesting small but statistically significant increased risk for secondary malignancy due to the cumulative dose of radiation exposure associated with diagnostic imaging. Children are most sensitive to radiation long term adverse effects. Therefore current pilot study will accrue adults only. If the result of this study will indicate potential advantage of PET-CT, this data can be weighted against radiation exposure risks to decide upon imaging strategies in pediatric patients with melanoma.

Exclusion Criteria:

1. Regional disease limited to an involved sentinel lymph node (occult or microscopic regional nodal metastasis).
2. Availability of prior PET-CT, performed within 60 days of initial clinical appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals over 18 years of age with metastatic melanoma (melanoma that has spread to other parts of the body) and are considered a candidate for surgery based on a contrast-enhanced computer tomography (CT) scan.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Percent of patients in whom a change in surgical plan occurred based on PET-CT result | Evaluation following PET-CT performed within 30 days of contrast-enhanced CT.

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Bronstein, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org